CLINICAL TRIAL: NCT02724865
Title: A Comparison Between Two Different Oral Appliance Therapies: Somnodent vs Herbst Appliance in Patients With Mild and Moderate OSA
Brief Title: Somnodent vs Herbst in Mild and Moderate OSA Patients
Acronym: COSH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, M.H.T. de Ruiter, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL44085.018.13
Record Dates: First submitted 2016-03-14; First posted 2016-03-31 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Oral Appliance Therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral appliance therapy; Somnodent® (Active Comparator): Somnodent is a duobloc appliance, which is frequently used in OSA treatment and is titratable.
  Interventions: Device: Somnodent® (Oral appliance therapy)
- Oral appliance therapy; Herbst® (Active Comparator): Herbst is a duobloc appliance, which is frequently used in OSA treatment and is titratable.
  Interventions: Device: Herbst® (Oral appliance therapy)

INTERVENTIONS:
Device: Somnodent® (Oral appliance therapy)
  Arms: Oral appliance therapy; Somnodent®
Device: Herbst® (Oral appliance therapy)
  Arms: Oral appliance therapy; Herbst®

SUMMARY:
Obstructive sleep apnea (OSA) is a common chronic sleep disorder that often requires lifelong care. The prevalence in the Netherlands is estimated around 300.000 patients. Due to longer life expectancy and increase in weight in the general population, its prevalence is expected to rise. Patients with mild and moderate OSA are treated primarily with an oral appliance at present time. Different oral appliances are available, but most used is the mandibular advancement device (MAD). This study focuses on two different types of MAD: the classic Herbst appliance, which is attached to the mandible and the maxilla and has an iron bar to regulate the open space; and the Somnodent, which consists of two separate splints, fixed on the mandible and the maxilla, but has no iron bar attached.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Ability to speak, read, and write Dutch.
* Ability to follow-up.
* Ability to use a computer with internet connection for online questionnaires.
* Diagnosis with symptomatic mild or moderate OSA (5 < AHI < 30).
* Expected to maintain current lifestyle (sports, medicine, diet, etc.)

Exclusion Criteria:

* Untreated periodontal problems, dental pain, and a lack of retention possibilities for an MAD.
* Medication used/related to sleeping disorders.
* Evidence of respiratory/sleep disorders other than OSA (eg. central sleep apnea syndrome).
* Systemic disorders (based on medical history and examination; e.g. rheumatoid arthritis)
* Temporomandibular disorders (based on the function examination of the masticatory system).
* Medical history of known causes of tiredness by day, or severe sleep disruption (insomnia, Periodic Limb Movement Disorder, Narcolepsy).
* Known medical history of mental retardation, memory disorders, or psychiatric disorders.
* Reversible morphological upper airway abnormalities (e.g. enlarged tonsils). - Inability to provide informed consent.
* simultaneous use of other modalities to treat OSA.
* Previous treatment with a MAD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypnea-Index (AHI) | 12 months
  AHI is measured with polysomnography in hospital
Oxygen-desaturation-Index | 12 months
  ODI is measured with polysomnography in hospital

SECONDARY OUTCOMES:
Epworth Sleeping Scale | 12 months
  Questionnaire
Functional Outcome of Sleep Questionnaire | 12 months
  Questionnaire
Blood pressure | 12 months
  physical examination
Euroqol (EQ-5D-3L) | 12 months
  Questionnaire

OTHER OUTCOMES:
Heart Rate | 12 months
  physical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Background] Young TB. Epidemiology of daytime sleepiness: definitions, symptomatology, and prevalence. J Clin Psychiatry. 2004;65 Suppl 16:12-6. PMID 15575799
- [Result] Hoekema A, Stegenga B, De Bont LG. Efficacy and co-morbidity of oral appliances in the treatment of obstructive sleep apnea-hypopnea: a systematic review. Crit Rev Oral Biol Med. 2004 Jun 4;15(3):137-55. doi: 10.1177/154411130401500303. PMID 15187032
- [Derived] Shi X, Lobbezoo F, Chen H, Rosenmoller BRAM, Berkhout E, de Lange J, Aarab G. Effects of mandibular advancement devices on upper airway dimensions in obstructive sleep apnea: responders versus non-responders. Clin Oral Investig. 2023 Sep;27(9):5649-5660. doi: 10.1007/s00784-023-05186-w. Epub 2023 Aug 17. PMID 37589748
- [Derived] Shi X, Lobbezoo F, Chen H, Rosenmoller BRAM, Berkhout E, de Lange J, Aarab G. Comparisons of the effects of two types of titratable mandibular advancement devices on respiratory parameters and upper airway dimensions in patients with obstructive sleep apnea: a randomized controlled trial. Clin Oral Investig. 2023 May;27(5):2013-2025. doi: 10.1007/s00784-023-04945-z. Epub 2023 Mar 17. PMID 36928350